CLINICAL TRIAL: NCT04385511
Title: Feasibility of Preoxygenation by Supraglottic Jet Ventilation Substituted for Mask Pressurized Ventilation Before Endotracheal Intubation:A Randomized Controlled Trail
Brief Title: Feasibility of Preoxygenation by Supraglottic Jet Ventilation Before Endotracheal Intubation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Hansheng Liang, Principal Investigator, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020PHB014-01
Record Dates: First submitted 2020-03-24; First posted 2020-05-13 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Preoxygenation
Keywords: jet ventilation; supraglottic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- supraglottic jet ventilation group (Experimental): Check blood gas before induction without preoxygen. Take stomach-ultrasound. Induction with Midazolam 0.02 mg/kg, sufentanil 0.3 ~ 0.5 ug/kg, propofol 2-2.5 mg/kg, rocuronium 0.6 mg/kg.After patients fall asleep and can't be woke up ,the investigators will put the Wei NASAL JET（WNJ）into one's nose to give the supraglottic jet ventilation with the driving pressure 0.01-0.03 megapascal (MPa), respiratory rate 15 beats per minute（BPM）, inspiratory/expiratory rate 1-1. 5.Check blood gas,stomach-ultrasound after 3 min, then do the tracheal intubation guided by visual laryngoscope.Stop jet ventilation during intubation.
  Interventions: Device: supraglottic jet ventilation
- mask pressurized ventilation group (No Intervention): Check blood gas before induction without preoxygen. Take stomach-ultrasound. Induction with Midazolam 0.02 mg/kg, sufentanil 0.3 ~ 0.5 ug/kg, propofol 2-2.5 mg/kg, rocuronium 0.6 mg/kg.After patients fall asleep and can't be woke up ,the investigators will give them 1 min mask pressure respiration, by pressure control "V - E technique" after muscle relaxant. Check blood gas,stomach-ultrasound after 2 min, then do the tracheal intubation guided by visual laryngoscope.

INTERVENTIONS:
Device: supraglottic jet ventilation — patients who were randomized into supraglottic jet ventilation group would be placed Wei Nasal Jet Tube after conducted. Then they will get the supraglottic jet ventilation to make sure their pulse oximetry is over 95%. After 3 minutes, endotracheal intubation was performed via mouth approach.
  Arms: supraglottic jet ventilation group

SUMMARY:
The study assumed that supraglottic jet ventilation is an alternative solution as a safe way to do the preoxygenation before endotracheal intubation by contrasting it with mask pressurized ventilation. The investigators also expected that supraglottic jet ventilation won't increase the occurrence of esophageal reflux.

DETAILED DESCRIPTION:
The study assumed that supraglottic jet ventilation is an alternative solution as a safe way to do the preoxygenation before endotracheal intubation by contrasting it with mask pressurized ventilation. The investigators also expected that supraglottic jet ventilation won't increase the occurrence of esophageal reflux.

The investigators randomly divided the patients into 2 groups:Group C and Group S.Patients in Group C will be preoxygenation with mask pressurized ventilation while patients in Group S with supraglottic jet ventilation by Wei NASAL JET（WNJ）.The tracheal intubation will be done after the 3 minutes preoxygenation. The investigators will measure the PaCO2 before and after preoxygenation, and the investigators will take the stomach-ultrasonography to find if there are too much gas in the gastro. If pulse oximetry is lower than 95% during the preoxygenation, the investigators will adjust the position of the Wei NASAL JET（WNJ) or use the change the way that the investigators hold the mask or change the pressure of ventilation on the basis of the group.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for any surgery under general anesthesia
* adults age range from 18-64 years old
* American Society of Anesthesiologists Physical Status Classification (ASA class) I-II
* voluntary participation in this clinical trail, signed informed consents

Exclusion Criteria:

* patients with epistaxis, rhinostenosis, the episodes of rhinitis, severe gastroesophageal reflux disease, severe respiratory disease, severe cardiovascular and cerebrovascular disease
* long-term use if anticoagulant drugs
* can't cooperate with intervention
* pulse oximetry <95% with normal respiration

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
alveolar oxygen tension（PaO2） | 3 minutes after preoxygenation
  The results comes from blood gas analysis
alveolar oxygen tension（PaO2） | baseline (before preoxygenation)
  The results comes from blood gas analysis

SECONDARY OUTCOMES:
PaCO2 | 3 minutes after preoxygenation
  The results comes from blood gas analysis
PaCO2 | baseline (before preoxygenation)
  The results comes from blood gas analysis
gastric antrum cross section | 3 minutes after preoxygenation
  The results comes from the ultrasound of gastric
gastric antrum cross section | baseline (before preoxygenation)
  The results comes from the ultrasound of gastric
complications | 1 day
  such as nasal bleeding, dry throat itching, sore throat, nausea and vomiting, pressure and other adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Hansheng Liang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China